CLINICAL TRIAL: NCT04664465
Title: PRediction of DIverse Glucocorticoids ToxIcity OUtcomeS
Acronym: PRODIGIOUS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0274
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Rheumatism; Polymyalgia Rheumatica; Giant Cell Arteritis; Idiopathic Inflammatory Myopathies; ANCA Associated Vasculitis; Systemic Autoimmune Disease
MeSH Terms: conditions — Rheumatic Fever; Polymyalgia Rheumatica; Giant Cell Arteritis; Myositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To date, there is no available tool that allows, at individual level, determination of the probability to develop clinically relevant complications of prolonged glucocorticoid therapy. In patients with inflammatory rheumatic disorders requiring prolonged glucocorticoid therapy, such tool could be useful to adapt first-line treatment decisions (in daily practice and in future clinical trials). The main objective of the study is to identify routine clinical, biological and DXA baseline characteristics predictive of the occurrence of clinically relevant complications of glucocorticoid therapy at 1 year, in order to propose a predictive score.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 1 year.
* Indication to initiate prolonged glucocorticoid therapy at a dosage ≥ 15 mg/day for the treatment of an inflammatory rheumatic disease.
* Initial treatment or relapse.
* Previsional treatment duration > 3 months.

Exclusion Criteria:

* Unable to consent.
* Previous corticosteroid therapy in the last 3 months at a significant dosage (> 5 mg per day).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients usually treated with prolonged glucocorticoid therapy in the field of rheumatology.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant complication of glucocorticoid therapy | 1 year
  The occurrence of one or more clinically relevant complication of glucocorticoid therapy during the first year of treatment, according to the Glucocorticoid Toxicity Index (items and specific list).

SECONDARY OUTCOMES:
Quality of life assessed through SF-36 | 1 year

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU d'Angers, Angers
  - CHRU de Brest, Brest
  - CHD Vendée, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CH des Pays de Morlaix, Morlaix
  - CHU de Nantes, Nantes
  - CHR d'Orléans, Orléans
  - <CHU de Poitiers, Poitiers
  - CHIC Quimper, Quimper
  - Clinique St Exupéry, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.